CLINICAL TRIAL: NCT00787254
Title: A Study to Investigate the Preventive Effect of AG-1749 Against the Recurrence of Gastric and Duodenal Ulcers During Long-term Treatment With Nonsteroid Anti-inflammatory Drug
Brief Title: Efficacy and Safety of Lansoprazole on Gastric and Duodenal Ulcers in Patients Taking Nonsteroidal Anti-Inflammatory Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-1749-CCT-352; 070495 (Registry Identifier: JapicCTI); U1111-1114-2071 (Registry Identifier: WHO); R100126 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Stomach Ulcer; Duodenal Ulcer
Keywords: Curling Ulcer; Gastric Ulcer; Nonsteroid anti-inflammatory drug; Drug Therapy
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole; Gefarnate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lansoprazole 15 mg QD (Experimental)
  Interventions: Drug: Lansoprazole
- Gefarnate 50 mg BID (Active Comparator)
  Interventions: Drug: Gefarnate

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 15 mg, capsules, orally, once daily and gefarnate placebo-matching capsules, orally, twice daily for up to 6 to 24 months.
  Other Names: AG-1749
  Arms: Lansoprazole 15 mg QD
Drug: Gefarnate — Gefarnate 50 mg, capsules, orally, twice daily and lansoprazole placebo-matching capsules, orally, once daily for up to 6 to 24 months.
  Arms: Gefarnate 50 mg BID

SUMMARY:
The purpose of this study is to determine whether AG-1749 (lansoprazole), once daily (QD), is effective in preventing the recurrence of gastric and duodenal ulcers in patients receiving long term treatment with nonsteroid anti-inflammatory drug, compared to gefarnate, twice daily (BID).

DETAILED DESCRIPTION:
In Japan, nonsteroid anti-inflammatory drug is one of common prescribed drugs for patients as an analgesic antipyretic, treating symptoms of cold, antiphlogistic and management of pain with rheumatoid arthritis, osteoarthrosis, lumbago. On the other hand, this nonsteroid anti-inflammatory drug sometimes causes gastric and duodenal ulcers and this ulcer leads to the gastrointestinal bleeding which may be cause of death.

The purpose of this study is to assess the efficacy of lansoprazole versus gefarnate in patients with a history of gastric or duodenal ulcers receiving daily nonsteroid anti-inflammatory medication.

ELIGIBILITY:
Inclusion Criteria:

* The patient was on nonsteroid anti-inflammatory drug (NSAID) treatment on the day when consent was obtained, and requires the long-term continuous treatment even after treatment with the investigational drug is started.
* The patient was confirmed to have a history of gastric ulcer or duodenal ulcer.

Exclusion Criteria:

* Endoscopically confirmed gastric and/or duodenal ulcers on Day 1.
* Endoscopically confirmed active upper gastrointestinal hemorrhage on Day 1.
* Current or past history of aspirin-induced asthma or hypersensitivity to NSAIDs.
* Past or planned surgery affecting gastric acid secretion.
* Clinically significant hepatic or renal disorder.
* Serious cardiac dysfunction, hypertension, or hematological disorder.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (68):
- Japan (68):
  - Kasugai-shi, Aichi-ken
  - Yotsukaido-shi, Chiba
  - Matsuyama, Ehime
  - Fukui-shi, Fukui
  - Chikushi-gun, Fukuoka
  - Fukuoka, Fukuoka
  - Kurume-shi, Fukuoka
  - Munakata-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Gifu, Gifu
  - Maebashi, Gunma
  - Higashihiroshima-shi, Hiroshima
  - Kure-shi, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Chitose-shi, Hokkaido
  - Sapporo, Hokkaido
  - Kato-shi, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Hitachi-Naka, Ibaraki
  - Yuki-shi, Ibaraki
  - Hakusan-shi, Ishikawa-ken
  - Komatsu-shi, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yamato-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Susaki-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Ise-shi, Mie-ken
  - Shima-shi, Mie-ken
  - Yokkaichi-shi, Mie-ken
  - Sendai, Miyagi
  - Ebino-shi, Miyazaki
  - Miyazaki, Miyazaki
  - Miyazaki-gun, Miyazaki
  - Matsumoto-shi, Nagano
  - Omura-shi, Nagasaki
  - Niigata, Niigata
  - Beppu-shi, Oita Prefecture
  - Okayama, Okayama-ken
  - Daito-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Ogi-shi, Saga-ken
  - Saga, Saga-ken
  - Hanyu-shi, Saitama
  - Sunto-gun, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Naruto-shi, Tokushima
  - Tokushima, Tokushima
  - Chuo-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Kiyose-shi, Tokyo
  - Machida-shi, Tokyo
  - Meguro-ku, Tokyo
  - Nishi-Tokyo-shi, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toshima-ku, Tokyo
  - Tottori-shi, Tottori
  - Yonago-shi, Tottori
  - Shimonoseki-shi, Yamaguchi
  - Yanai-shi, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at sites in Japan from April 2007 to May 2009.
Pre-assignment Details: Participants were enrolled in either lansoprazole, once daily (QD) or gefarnate, twice daily (BID) treatment groups. NSAID = Nonsteroidal anti-inflammatory drug.
Groups:
- Lansoprazole 15 mg QD: Lansoprazole 15 mg, capsules, orally, once daily and gefarnate placebo-matching capsules, orally, twice daily for up to 6 to 24 months.
- Gefarnate 50 mg BID: Gefarnate 50 mg, capsules, orally, twice daily and lansoprazole placebo-matching capsules, orally, once daily for up to 6 to 24 months.
Period: Overall Study
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Started | 185 | 181
Completed | 109 | 99
Not Completed | 76 | 82
Not completed — Adverse Event | 24 | 23
Not completed — Protocol Violation | 26 | 23
Not completed — Withdrawal by Subject | 16 | 11
Not completed — Lack of Efficacy | 4 | 15
Not completed — NSAIDs discontinuation | 1 | 2
Not completed — Institution closed | 1 | 0
Not completed — Physician Decision | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID | Total
Number analyzed (Participants) | 185 | 181 | 366
Age, Customized [Number; unit: participants]
  ≤39 years | 7 (3.8) | 6 (3.3) | 13 (3.6)
  Between 40 and 49 years | 18 (9.7) | 13 (7.2) | 31 (8.5)
  Between 50 and 59 years | 38 (20.5) | 43 (23.8) | 81 (22.1)
  Between 60 and 64 years | 33 (17.8) | 29 (16.0) | 62 (16.9)
  Between 65 and 69 years | 33 (17.8) | 30 (16.6) | 63 (17.2)
  Between 70 and 79 years | 43 (23.2) | 48 (26.5) | 91 (24.9)
  ≤80 years | 13 (7.0) | 12 (6.6) | 25 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 107 | 219
  Male | 73 | 74 | 147
Region of Enrollment [Number; unit: participants]
  Japan | 185 | 181 | 366

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastric Ulcer and/or Duodenal Ulcer
Description: The number of participants that developed gastric ulcer and/or duodenal ulcer at month 24 or final visit. Ulcers are defined as mucosal defect with white coating 3 mm or greater.
Time Frame: 24 Months
Population: Participants not taking investigational drug were not included.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 183 | 181
participants | 15 | 46
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.2510, 95% CI 2-sided [0.1400 to 0.4499]

2. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 3)
Description: The Lanza score (partially revised) attributes the severity of induced erosive mucosal injury in the stomach, graded on a 5 point scale (0=normal; 1= erosion/hemorrhage in one area of the stomach and <1 lesion; 2= erosion/hemorrhage in one area of the stomach with 2-5 lesions; 3= erosion/hemorrhage in two areas in the stomach/one area involves >6 lesions; 4= erosion/hemorrhage appear in three or more areas in the stomach). Erosions are mucosal defect < 3 mm. Ulcers are mucosal defect with white coating ≥ 3 mm. Higher scores indicate greater severity of gastric mucosal injury.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 167 | 154
scores on a scale | -0.114 (1.020) | 0.429 (1.318)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 6)
Description: as for outcome 2
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 116 | 85
scores on a scale | -0.319 (1.060) | 0.188 (1.268)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0041, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 12)
Description: as for outcome 2
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 78 | 62
scores on a scale | -0.231 (1.299) | 0.048 (1.137)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0652, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 18)
Description: as for outcome 2
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 37 | 18
scores on a scale | -0.162 (1.280) | -0.278 (1.227)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.9836, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 24)
Description: as for outcome 2
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 5 | 2
scores on a scale | -0.800 (1.304) | NA (NA) — No test was performed when the number of cases was 5 or less.

7. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 3)
Description: The Lanza score (partially revised) attributes the severity of induced erosive mucosal injury in the duodenum, graded on a 4 point scale (0=normal; 1= erosion and hemorrhage are localized in one area of the duodenum and < 1 lesion; 2= 2 to 5 lesions ; 3= > 6 lesions). Erosions are defined as mucosal defect < 3 mm. Ulcers are defined as mucosal defect with white coating ≥ 3 mm. Higher scores indicate greater severity of duodenal mucosal injury.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 167 | 155
scores on a scale | -0.102 (0.499) | 0.142 (0.649)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 6)
Description: as for outcome 7
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 116 | 86
scores on a scale | -0.095 (0.527) | 0.047 (0.373)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0161, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 12)
Description: as for outcome 7
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 79 | 62
scores on a scale | -0.177 (0.675) | 0.048 (0.381)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0068, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 18)
Description: as for outcome 7
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 37 | 18
scores on a scale | -0.297 (0.812) | -0.056 (0.539)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2363, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 24)
Description: as for outcome 7
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 5 | 2
scores on a scale | -0.200 (0.447) | NA (NA) — No test was performed when the number of cases was 5 or less.

12. Secondary Outcome: Number of Participants With Gastric or Duodenal Ulcer or Gastric or Duodenal Hemorrhagic Lesion (Upper Gastrointestinal Hemorrhage)
Description: Number of participants with gastric or duodenal ulcer or gastric or duodenal hemorrhagic lesion (upper gastrointestinal hemorrhage) from baseline through month 24 or final visit. Ulcers are defined as mucosal defect with white coating 3 mm or greater.
Time Frame: On occurrence (up to month 24).
Population: On days where participants did not have an occurrence of gastric or duodenal ulcer or gastric or duodenal hemorrhagic lesion (upper gastrointestinal hemorrhage) and who also underwent endoscopic examination were considered censored dates. Values are from the Full Analysis Set.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 183 | 181
participants | 15 | 52
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Log Rank

13. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop postprandial pain at month 3, and number of participants that develop postprandial pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | -0.006 (0.178) | 0.014 (0.319)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4788, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop postprandial pain at month 6, and number of participants that develop postprandial pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.027 (0.285) | 0.000 (0.347)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.6607, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop postprandial pain at month 12, and number of participants that develop postprandial pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | -0.014 (0.208) | -0.020 (0.249)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8811, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop postprandial pain at month 18, and number of participants that develop postprandial pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | 0.000 (0.000) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop postprandial pain at month 24, and number of participants that develop postprandial pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

18. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop hunger and nighttime pain at month 3, and number of participants that develop hunger and nighttime pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | -0.044 (0.326) | 0.014 (0.400)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2060, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop hunger and nighttime pain at month 6, and number of participants that develop hunger and nighttime pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.009 (0.393) | -0.036 (0.424)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.5099, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop hunger and nighttime pain at month 12, and number of participants that develop hunger and nighttime pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | -0.029 (0.416) | -0.061 (0.317)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7794, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop hunger and nighttime pain at month 18, and number of participants that develop hunger and nighttime pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | 0.000 (0.000) | 0.000 (0.447)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop hunger and nighttime pain at month 24, and number of participants that develop hunger and nighttime pain at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

23. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop the feeling of an enlarged abdomen at month 3, and number of participants that develop the feeling of an enlarged abdomen at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | -0.025 (0.318) | -0.014 (0.452)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.6980, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop the feeling of an enlarged abdomen at month 6, and number of participants that develop the feeling of an enlarged abdomen at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.000 (0.381) | -0.048 (0.408)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4599, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop the feeling of an enlarged abdomen at month 12, and number of participants that develop the feeling of an enlarged abdomen at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | -0.057 (0.336) | -0.204 (0.407)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0355, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop the feeling of an enlarged abdomen at month 18, and number of participants that develop the feeling of an enlarged abdomen at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | -0.056 (0.416) | 0.000 (0.447)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7325, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop the feeling of an enlarged abdomen at month 24, and number of participants that develop the feeling of an enlarged abdomen at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

28. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop the feeling of nausea at month 3, and number of participants that develop the feeling of nausea at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | -0.006 (0.239) | 0.007 (0.308)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8262, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop the feeling of nausea at month 6, and number of participants that develop the feeling of nausea at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.009 (0.286) | -0.012 (0.245)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7244, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop the feeling of nausea at month 12, and number of participants that develop the feeling of nausea at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | -0.043 (0.204) | -0.041 (0.200)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.9566, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop the feeling of nausea at month 18, and number of participants that develop the feeling of nausea at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | 0.000 (0.000) | -0.091 (0.302)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2008, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop the feeling of nausea at month 24, and number of participants that develop the feeling of nausea at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

33. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop the feeling of heartburn at month 3, and number of participants that develop the feeling of heartburn at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | -0.057 (0.378) | 0.058 (0.625)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0703, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop the feeling of heartburn at month 6, and number of participants that develop the feeling of heartburn at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | -0.027 (0.476) | -0.095 (0.428)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.3046, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop the feeling of heartburn at month 12, and number of participants that develop the feeling of heartburn at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | -0.114 (0.363) | -0.102 (0.510)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7121, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop the feeling of heartburn at month 18, and number of participants that develop the feeling of heartburn at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | -0.056 (0.236) | 0.091 (0.302)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.1522, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop the feeling of heartburn at month 24, and number of participants that develop the feeling of heartburn at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | -1.000 (NA) — No test was performed when the number of cases was 5 or less. |

38. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 3)
Description: The number of participants that develop anorexia at month 3, and number of participants that develop anorexia at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | 0.006 (0.138) | 0.022 (0.283)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.5328, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 6)
Description: The number of participants that develop anorexia at month 6, and number of participants that develop anorexia at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.036 (0.187) | 0.024 (0.268)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7223, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 12)
Description: The number of participants that develop anorexia at month 12, and number of participants that develop anorexia at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | 0.014 (0.208) | -0.020 (0.143)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.3117, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 18)
Description: The number of participants that develop anorexia at month 18, and number of participants that develop anorexia at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | 0.056 (0.236) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4344, t-test, 2 sided

42. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 24)
Description: The number of participants that develop anorexia at month 24, and number of participants that develop anorexia at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

43. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 3)
Description: The number of participants that experience hematemesis and melena (blood stool, black stool, tarry stool) at month 3, and number of participants that experience hematemesis and melena at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 138
scores on a scale | 0.006 (0.080) | -0.007 (0.085)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.1571, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 6)
Description: The number of participants that experience hematemesis and melena (blood stool, black stool, tarry stool) at month 6, and number of participants that experience hematemesis and melena at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 84
scores on a scale | 0.000 (0.000) | 0.012 (0.109)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2503, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 12)
Description: The number of participants that experience hematemesis and melena (blood stool, black stool, tarry stool) at month 12, and number of participants that experience hematemesis and melena at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 70 | 49
scores on a scale | 0.043 (0.359) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4028, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 18)
Description: The number of participants that experience hematemesis and melena (blood stool, black stool, tarry stool) at month 18, and number of participants that experience hematemesis and melena at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 18.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 18 | 11
scores on a scale | 0.000 (0.000) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney)

47. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 24)
Description: The number of participants that experience hematemesis and melena (blood stool, black stool, tarry stool) at month 24, and number of participants that experience hematemesis and melena at baseline. It is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 24.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 1 | 0
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. |

48. Secondary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug. A TEAE may also be a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing. Please see Other Adverse Events table below for TEAE listings.
Time Frame: Per Incidence (up to 24 months).
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 183 | 181
participants
  Adverse Event | 154 | 125
  Adverse event (Frequency ≥5%) | 83 | 64
  Adverse event related to the study drug | 28 | 28
  Serious adverse event | 29 | 17
  Serious adverse event related to the study drug | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were summarized by onset date occurring on or after the first dose of double-blind study medication, and up to 24 months after the permanent discontinuation of the double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Serious Adverse Events (participants affected / at risk) | 29/183 | 17/181
Other Adverse Events (participants affected / at risk) | 83/183 | 64/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg QD (N=183) | Gefarnate 50 mg BID (N=181)
Colonic polyp (Gastrointestinal disorders) | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Collagen disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 1
Medical device pain (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg QD (N=183) | Gefarnate 50 mg BID (N=181)
Nasopharyngitis (Infections and infestations) | 51 | 37
Diarrhea (Gastrointestinal disorders) | 19 | 5
Reflux esophagitis (Gastrointestinal disorders) | 4 | 12
Constipation (Gastrointestinal disorders) | 10 | 10
Fall (Injury, poisoning and procedural complications) | 12 | 10
Eczema (Skin and subcutaneous tissue disorders) | 10 | 5

LIMITATIONS AND CAVEATS:
This study was prematurely discontinued due to results available from a parallel study (AG-1749-CCT-351; NCT00762359) demonstrating a preventive effect on ulcer occurrence which impacted the risk/benefit profile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.